CLINICAL TRIAL: NCT03605420
Title: Effects of the Visit Prior to Hospital Admission on Anxiety, Depression and Satisfaction of Family in an Intensive Care Unit
Brief Title: Relatives Visit Prior to Hospital Admission & Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de León (Other)
Responsible Party: Principal Investigator, César Calvo Lobo, PhD, MSc, PT, Universidad de León
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: ICU-visit-relatives
Record Dates: First submitted 2018-07-21; First posted 2018-07-30 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Anxiety; Depression; Care Unit Syndrome
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Receiving one family visit prior to hospital admission
  Interventions: Other: Family visit prior to hospital admission
- Control group (No Intervention): Without receiving one family visit prior to hospital admission

INTERVENTIONS:
Other: Family visit prior to hospital admission — Family receiving one visit prior to hospital admission for surgery
  Arms: Experimental group

SUMMARY:
The present study evaluates the effects of the visit prior to hospital admission on anxiety, depression and satisfaction of family in an intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Family of a patient for hospital admission for surgery

Exclusion Criteria:

* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
The Hospital Anxiety and Depression Scale | Change from Baseline anxiety and depression at 90 days
  Anxiety subscale range from 0 to 21. Depression subscale range from 0 to 21. Higher values represent a worse outcome (higher depression or anxiety).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital La Princesa, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided